CLINICAL TRIAL: NCT03055416
Title: Mobile Phone Intervention for Physical Activity Maintenance in African American Men (MobileMen) Ph I
Brief Title: Mobile Phone Intervention for Physical Activity Maintenance in African American Men (MobileMen)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: Pennington Biomedical Research Center (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0312; 1R41MD010304-01A1 (NIH)
Record Dates: First submitted 2017-01-16; First posted 2017-02-16 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Overweight and Obesity
Keywords: Overweight; Obesity; Physical Activity; African-American Men; mHealth; Mobile Health
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mobile Men App Prototype (Other): Prototype of physical activity mobile app geared for African-American men.
  Interventions: Other: Mobile Men App Prototype

INTERVENTIONS:
Other: Mobile Men App Prototype — Testing of app functionality

SUMMARY:
African American men are at risk of developing chronic disease partly due to low levels of regular physical activity. Studies have been effective in increasing physical activity levels in African American men; however for the health benefits of exercise to be maintained continued physical activity is necessary. The purpose of the current study is to develop a mobile phone application for African American men that will help them maintain their physical activity levels.

DETAILED DESCRIPTION:
African American men experience health disparities across a number of preventable chronic diseases, including cardiovascular disease, strokes, obesity, and diabetes. Physical activity (PA) is a modifiable risk factor for these conditions. The few PA promotion studies that have included African American men have resulted in successful short-term behavior change, yet in order for the health benefits of PA to be realized, PA levels must be maintained. While behavior change maintenance programs have been shown to assist participants in sustaining behavior change, we were unable to identify any studies that have developed maintenance programs specifically targeting African American men. The purpose of this proposal is to develop a PA maintenance program for African American men. This Phase I Small Business Technology Transfer (STTR) project, MobileMen, will deliver the intervention utilizing mobile health (mHealth) technology and therefore, will be led by researchers and multimedia developers at Klein Buendel, Inc. (KB) and Pennington Biomedical Research Center (Dr. Newton, PI). The use of mHealth, as opposed to other avenues of intervention delivery, is based on published reports documenting that African Americans perceive mobile technology as an acceptable means of intervention delivery. In addition, ownership of smartphones and the use of text messaging are highest among African Americans compared to other ethnic groups. There is a need to tailor this intervention towards African American men because they have unique gender role beliefs which influence exercise promotion. There is also increasing recognition of the need for researchers to develop interventions in collaboration with the target population. Therefore, the current proposal will involve conducting formative research with African American men to identify the key elements for program development. The fact that mHealth is acceptable to- and the fact that the application will be developed in collaboration with African American men, leads us to hypothesize that African American men will view the mHealth intervention as acceptable, feasible, and usable. In this Phase I STTR, KB will: (1) conduct multi-method formative research to guide app design and content, (2) produce a functioning app prototype, and (3) conduct usability testing on the prototype for functionality, ease of use, and interest among African American men. To KB's knowledge, no study has utilized mobile phones as a means of effecting PA levels in African American men. MobileMen will address an unmet need in the marketplace as it will be the first smartphone app that is targeted toward PA maintenance in African American men.

ELIGIBILITY:
Inclusion Criteria:

* Owns a smartphone and speaks and reads English, lives in the Greater Baton Rouge area, and consents to participate.

Exclusion Criteria:

* Cognitive impairment that would interfere with participating in a group discussion, unwilling to be audio and video-recorded, or unwilling to give written informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2016-09; Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
System Usability Questionnaire | 5 months
  Participant perspective of program feasibility and physical activity promotion.

SECONDARY OUTCOMES:
User Perspectives Survey | 5 months
  Participant perspective of app's design and identifying and correcting usability problems.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Newton, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (2):
- United States (2):
  - Klein Buendel, Inc., Golden, Colorado
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):e2-e220. doi: 10.1161/CIR.0b013e31823ac046. Epub 2011 Dec 15. No abstract available. PMID 22179539
- [Background] Cowie CC, Rust KF, Byrd-Holt DD, Gregg EW, Ford ES, Geiss LS, Bainbridge KE, Fradkin JE. Prevalence of diabetes and high risk for diabetes using A1C criteria in the U.S. population in 1988-2006. Diabetes Care. 2010 Mar;33(3):562-8. doi: 10.2337/dc09-1524. Epub 2010 Jan 12. PMID 20067953
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of obesity in the United States, 2009-2010. NCHS Data Brief. 2012 Jan;(82):1-8. PMID 22617494
- [Background] LaMonte MJ, Barlow CE, Jurca R, Kampert JB, Church TS, Blair SN. Cardiorespiratory fitness is inversely associated with the incidence of metabolic syndrome: a prospective study of men and women. Circulation. 2005 Jul 26;112(4):505-12. doi: 10.1161/CIRCULATIONAHA.104.503805. Epub 2005 Jul 11. PMID 16009797
- [Background] LaMonte MJ, Blair SN, Church TS. Physical activity and diabetes prevention. J Appl Physiol (1985). 2005 Sep;99(3):1205-13. doi: 10.1152/japplphysiol.00193.2005. PMID 16103523
- [Background] Newton RL Jr, Griffith DM, Kearney WB, Bennett GG. A systematic review of weight loss, physical activity and dietary interventions involving African American men. Obes Rev. 2014 Oct;15 Suppl 4:93-106. doi: 10.1111/obr.12209. PMID 25196408